CLINICAL TRIAL: NCT02687295
Title: Metabolic Risk Markers and Body Weight Are Decreased by Green-plant Supplementation in a Pilot Study With Overweight-to-obese Middle-aged Men.
Brief Title: Improvement of Metabolic Health After Thylakoid Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Eva-Lena Stenblom, M.D., Region Skane
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Gubbar-2010
Record Dates: First submitted 2016-02-10; First posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Metabolic Syndrome; Obesity
MeSH Terms: conditions — Metabolic Syndrome; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Placebo Comparator): Control group subjects received the same diet restriction intervention as treatment group. However, their food products did not contain any active component.
  Interventions: Other: Control
- Thylakoid group (Active Comparator): Thylakoid group subjects received the same diet restriction intervention as the control group. However, their food products did contain an active component in the form of thylakoid powder.
  Interventions: Dietary Supplement: Thylakoids

INTERVENTIONS:
Dietary Supplement: Thylakoids
  Other Names: Appethyl; Green-plant membranes
  Arms: Thylakoid group
Other: Control
  Other Names: Placebo
  Arms: Control group

SUMMARY:
Objective:

The purpose of this study was to investigate the possible effects of green-plant thylakoid supplementation to a restricted diet intervention study in overweight to obese men.

Methods:

Overweight-obese men (BMI 25 - 35) were treated to a 30 E% restricted diet for one month, followed by one month of stabilization. Then they were divided in two treatment arms of one month each; one thylakoid-enriched diet (n=10) and one control diet (n=10). Body measurements and blood samples were taken throughout the study.

DETAILED DESCRIPTION:
Twenty healthy, non-vegetarian, non-smoking Caucasian men were included in the study. Inclusion criteria: men aged 40 to 70 years with a BMI of 25 to 35. Exclusion criteria: Metabolic disturbances, bariatric surgery, recent diet, food allergies or treatment with antibiotics. The study protocol was approved by the Ethical Committee of Lund University, Sweden (#2006/361).

The trial consisted of three periods: 1) diet-restriction period (one month) 2) stabilizing period (one month) 3) diet-restriction period with supplementation of thylakoids or placebo (one month). The two weight-losing periods included strict diet recommendation with -30 energy % (E%), and macronutrient composition: 55-65 E% carbohydrates, 10-15 E% protein and 25-35 E% fat. Sixty minutes of low intensive exercise per day was also required.

During the stabilizing month participants were instructed to eat a healthy diet to be able to keep their achieved weight-loss.

Day 0, 28, 56 and 84 the participants arrived after 12-hour fasting for blood sampling and anthropometric measurements. The blood samples were analyzed for plasma-glucose, insulin, HbA1c, inflammation markers, cholecystokinin, ghrelin, total cholesterol, LDL-cholesterol, HDL-cholesterol, and triacylglycerol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, overweight, non-vegetarian, non-smoking

Exclusion Criteria:

* Medication for metabolic disturbances, previous bariatric surgery, diabetes, had been on diet or treated with antibiotics during last 3 months, food-allergies

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Body weight | 3 months

SECONDARY OUTCOMES:
Waist circumference | 3 months
Blood lipids | 3 months
  Total cholesterol, LDL, HDL and TAG are measured fasting every fourth week.
P-glucose and p-insulin | 3 months
  P-glucose, p-insulin and HbA1c are measured fasting every fourth week.
Inflammatory markers | 3 months
  CRP and TNF alpha are measured fasting every fourth week.
Appetite regulating hormones | 3 months
  Ghrelin and leptin are measured fasting every fourth week.

CONTACTS AND LOCATIONS:
Overall Officials: Eva-Lena Stenblom, M.D., Principal Investigator — Lund University, Region Skane

IPD SHARING:
Plan to Share IPD: No